CLINICAL TRIAL: NCT07356505
Title: Efficacy and Safety of Micra AV2 Transcatheter Pacing System
Acronym: EMAV2
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: s70117
Record Dates: First submitted 2026-01-12; First posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: AV Block Complete; AV Block-2Nd Degree-Type 1; AV Block
Keywords: leadless pacemaker; Micra AV; AV synchrony
MeSH Terms: conditions — Atrioventricular Block

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Micra AV (Experimental): All patients will receive a Micra AV2 leadless pacemaker
  Interventions: Device: Implant procedure of a Micra AV2 leadless pacemaker (Medtronic)

INTERVENTIONS:
Device: Implant procedure of a Micra AV2 leadless pacemaker (Medtronic) — All patients will be implanted with aMicra AV2 leadless pacemaker

SUMMARY:
A third generation, Micra AV2 is now available and proposes increased automaticity and improved AV synchrony algorithms based on computing model. The new algorithms permit the delivery of AV synchronous pacing, improving the automatic AV synchrony at faster heart rates between 80-100 bpm with a maximal upper tracking rate limit of 135 bpm (previously 115-120 bpm in the Micra AV1). Micra AV2 presents also a potential extended longevity of 15.6 years (increased by > 44% in comparison of Micra AV1). Up to now, no clinical study has evaluated the efficacy and safety of Micra AV2 in a real-world setting.

The focus of this study is to characterize chronic ambulatory AV synchrony in patients with high degree AV block and normal sinus rhythm implanted with a Micra AV2 as primary objective to evaluate AV synchrony during exercise as secondary objective.

DETAILED DESCRIPTION:
Prospective, single-arm, multi-centre clinical study to characterize the chronic efficacy and safety profile of CE approved and market released Micra AV2 A sample size of approximately 150 subjects implanted with a Micra AV2 is required to evaluate the different objectives. A minimal sample size of 50 subjects with persistent 3rd degree AVB and normal sinus node function is required to evaluate the ambulatory AV synchrony at 6-month follow-up.

Primary objective:

Characterize ambulatory AV synchrony in subjects with persistent third degree AV block and normal sinus node function at 6-month post Micra AV2 implant procedure

Secondary objective(s):

1. Characterize the AV synchrony and device behaviour during exercise in subjects with persistent third degree AV block and normal sinus node function at 6-month post implant procedure
2. Characterize the evolution of left ventricular function at 12-month post implant
3. Evaluate the efficacy of the 'Atrial Sensing Setup' at the end of the implant procedure
4. Long-term follow-up (3 years) to evaluate AV synchrony, need for system revision and complication rate including rate of pacing induced cardiomyopathy

ELIGIBILITY:
Inclusion Criteria:

1. Voluntary written informed consent of the participant or their legally authorized representative has been obtained prior to any screening procedures
2. At least 18 years of age at the time of signing the Informed Consent Form (ICF)
3. Participant will be implanted with a Micra AV2 for an approved indication for use
4. Participant with a history of any type of high-degree AV block
5. Participant is willing and able to comply the study protocol

Exclusion Criteria:

-1. Subject implanted with a Micra AV2 on a non-permanent basis (e.g. CIED infection) 2. Subject is pregnant (if required by local law, women of child-bearing potential must undergo a pregnancy test within seven days prior to Micra AV2 implant procedure) 3. Subject currently enrolled or planning to participate in a potentially confounding drug or device trial during the study.

4. Subject meets any exclusion criteria required by local law (age or other)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2026-01-12 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
AV synchrony at 6 months | 6 months follow-up
  AV synchrony will be computed on an individual heartbeat basis and is defined as met for paced or sensed ventricular beats that are within 300 ms following an ECG confirmed P-wave. This endpoint will be used for the primary objective , for the secondary objective #1 (AV synchrony during exercise at 6-month post-implant) and for the secondary objective #3 (evaluation of the AV synchrony following the automated atrial sensing setup)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospitals of Leuven, Leuven, Flemish Brabant, Belgium